CLINICAL TRIAL: NCT06129305
Title: Comparison of the Distance of the Erector Spina Muscle From the Skin at Different Thoracal Levels and Different posıtıons Under Ultrasonography
Brief Title: Erector Spina Muscle Distance From the Skin at Different Thoracal Elevations
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Muhammed Halit Satici, Specialist, Department of Anesthesiology, Konya City Hospital, M.D, Konya City Hospital
Other Study IDs: konya city hospital
Record Dates: First submitted 2023-08-14; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Pain, Postoperative; Pain, Back
Keywords: Erector spinae plane block; interfascial plan block.
MeSH Terms: conditions — Pain, Postoperative; Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Comparison of the distance of the Erector Spina muscle from the skin at different thoracal levels and different posıtıons under ultrasonography — Comparison of the distance of the Erector Spina muscle from the skin at different thoracal levels and different posıtıons under ultrasonography

SUMMARY:
In our study, we aimed to calculate the ideal measurement of the distance of the erector spina muscle to the skin and to find the best ultrasonography image at different thoracic levels (T1-T2, T5-T6, T5-T6, T11-T12) and in other positions (lateral-sitting-pron) to improve the quality of the block in patients who will undergo erector spina plan block.

Our primary goal is to determine which thoracic level the erector spinae muscle is closer to the skin and whether the USG screen image is better. Our secondary goal is to find out in which position the erector spinae muscle is closer to the skin and the USG screen image is better.

DETAILED DESCRIPTION:
1- Abstract Introduction Erector spina plana block can be performed in different positions (sitting-lateral-pron) and at different thoracic levels. In our study, we aimed to calculate the ideal measurement of the distance of the erector spina muscle to the skin and to find the best ultrasonography image at different thoracic levels (T1-T2, T5-T6, T5-T6, T11-T12) and in other positions (lateral-sitting-pron) to improve the quality of the block in patients who will undergo erector spina plan block. Material and Methods A total of 80 patients (40 females and 40 males, ASA I-II) aged 18-65 years were included in the study. The erector spinae muscle was determined at T1-T2, T5-T6, and T11-T12 levels and in lateral, sitting, and prone positions, respectively, with a high frequency 10-15 millihertz linear probe of ultrasound, The distance from the skin to the midline of the ultrasound screen was measured, and the best ultrasound screen image was recorded. Erector spina plan block, distance measurement, different positions, interfascial plan block.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-65 years ASA (American Society of Anaesthesiologists) I-II who were to undergo cholecystectomy who were to undergo mastectomy who were to undergo inguinal hernia who were to undergo thoracic surgery

Exclusion Criteria:

Patients in whom peripheral nerve block was contraindicated uncooperative patients disabled patients emergency cases patients with scoliosis pregnant and breastfeeding women patients with trauma incision scars in the measured area ASA III-IV-V group patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18-65 years with ASA (American Society of Anaesthesiologists) I-II patients
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
distance of the erector spinae muscle from the skin in millimeters | two years
  Our primary goal is to determine which thoracic level the erector spinae muscle is closer to the skin and whether the USG screen image is better.

SECONDARY OUTCOMES:
clarity of the erector spinae muscle in different positions | two years
  Our secondary goal is to find out in which position the erector spinae muscle is closer to the skin and the USG screen image is better.

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMED H SATICI, M.D., Principal Investigator — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We do not have such an opinion.